CLINICAL TRIAL: NCT07202494
Title: Integrating Metabolism, Connectivity, and Mesoscale Imaging at Ultra-high Field to Decipher Mechanisms of Resilience and Neurodegeneration in Neurological Diseases and Healthy Aging
Acronym: MESO7
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RCAPHM23_0203
Record Dates: First submitted 2025-05-07; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis; Neuromyelitis Optica Spectrum Disorders; Myelin Oligodendrocyte Glycoprotein Antibody-Associated Disease (MOGAD); Alzheimer Disease; Parkinson Disease; Amyotrophic Lateral Sclerosis (ALS); Temporal Lobe Epilepsy; Epilepsy; Mild Traumatic Brain Injury; Healthy Aging
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica; Myelin Oligodendrocyte Glycoprotein Antibody-Associated Disease; Alzheimer Disease; Parkinson Disease; Amyotrophic Lateral Sclerosis; Epilepsy, Temporal Lobe; Epilepsy; Brain Concussion | interventions — X-Rays; Functional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Healthy controls: (160 participants, split by age and sex)
  Interventions: Other: Imaging Techniques (MRI 3T & 7T, Functional, Structural, and Metabolic Imaging)
- Multiple Sclerosis
  Interventions: Other: Imaging Techniques (MRI 3T & 7T, Functional, Structural, and Metabolic Imaging)
- Neuromyelitis Optica Spectrum Disorder (NMOSD)
  Interventions: Other: Imaging Techniques (MRI 3T & 7T, Functional, Structural, and Metabolic Imaging)
- Myelin Oligodendrocyte Glycoprotein Antibody Disease (MOGAD)
  Interventions: Other: Imaging Techniques (MRI 3T & 7T, Functional, Structural, and Metabolic Imaging)
- Alzheimer's Disease
  Interventions: Other: Imaging Techniques (MRI 3T & 7T, Functional, Structural, and Metabolic Imaging)
- Parkinson's Disease
  Interventions: Other: Imaging Techniques (MRI 3T & 7T, Functional, Structural, and Metabolic Imaging)
- Amyotrophic Lateral Sclerosis (ALS)
  Interventions: Other: Imaging Techniques (MRI 3T & 7T, Functional, Structural, and Metabolic Imaging)
- Temporal Epilepsy
  Interventions: Other: Imaging Techniques (MRI 3T & 7T, Functional, Structural, and Metabolic Imaging)
- Non-Temporal Epilepsy
  Interventions: Other: Imaging Techniques (MRI 3T & 7T, Functional, Structural, and Metabolic Imaging)
- Mild Traumatic Brain Injury (mTBI)
  Interventions: Other: Imaging Techniques (MRI 3T & 7T, Functional, Structural, and Metabolic Imaging)

INTERVENTIONS:
Other: Imaging Techniques (MRI 3T & 7T, Functional, Structural, and Metabolic Imaging) — Functional MRI (fMRI) Diffusion Tensor Imaging (DTI) Sodium Imaging (23Na-MRI) Phosphorus Imaging (31P-MRI)

SUMMARY:
The MESO7 study is a prospective observational research project designed to investigate the mechanisms of resilience and neurodegeneration in neurological diseases and healthy aging. It leverages advanced multiparametric brain and spinal cord imaging at high (3T) and ultra-high magnetic fields (7T) to assess structural, functional, metabolic, and mesoscale changes in the central nervous system (CNS). Particular emphasis is placed on sodium (23Na-MRI) and phosphorus (31P-MRI) imaging, along with layer-dependent brain connectivity analysis.

The primary objective is to evaluate the impact of neuronal energy failure, measured via sodium concentration, on functional and structural reorganization in both healthy individuals and patients with various neurological conditions. Directed brain network models will be constructed from MRI data to quantify the connectivity strength (in- and out-degree) of cortical nodes. These connectivity metrics will be correlated with sodium concentrations to assess energy failure and its role in network reorganization. Longitudinal follow-up over two years is planned for subgroups with clinically progressive diseases.

Secondary objectives include decoding metabolic, microstructural, and functional signatures of successful aging at the laminar level; characterizing disease-specific patterns of cortical and spinal microstructure associated with physical and cognitive dysfunction; describing longitudinal mesoscale and metabolic changes; and generating representative normative imaging datasets for the neuroscience community.

The study plans to enroll a total of 540 patients across 9 neurological conditions:Multiple Sclerosis (MS), Neuromyelitis Optica Spectrum Disorders (NMOSD), MOG Antibody Disease (MOGAD), Alzheimer's disease, Parkinson's disease, Amyotrophic Lateral Sclerosis (ALS), temporal and non-temporal epilepsy, and mild traumatic brain injury (mTBI),in addition to 160 age- and sex-matched healthy controls, totaling 700 participants. Imaging and clinical assessments will be performed at the CEMEREM center at Timone University Hospital, AP-HM, Marseille, France.

Each participant will undergo multiparametric brain and spinal cord MRI, including DTI, BOLD, MP2RAGE, SWI, quantitative sodium and phosphorus imaging, and functional assessments including neuropsychological testing, visual and motor function tests. Disease-specific assessments such as OCT, evoked potentials, and disability scores (e.g., EDSS for MS) will also be included when appropriate.

The study is expected to improve understanding of CNS adaptation mechanisms and support the development of more accurate diagnostic and prognostic tools for neurodegenerative diseases

ELIGIBILITY:
Inclusion Criteria:

* Age:Female or male, aged 18 years or older.
* Health Status: No uncontrolled general diseases, such as cancer, autoimmune diseases, liver failure, severe or untreated high blood pressure, or severe rhythm disorders. No chronic psychiatric illnesses, including severe dementia.
* MRI Compatibility: No contraindications for MRI exams (e.g., claustrophobia, metal foreign bodies, pacemakers, severe kidney failure).
* Social Security Coverage: Participants must have social security coverage.
* Informed Consent: The participant must have read, understood, and signed the informed consent after being adequately informed about the study.
* Specific Disease Criteria (For Disease Groups): Specific inclusion criteria apply to each pathology, such as MS (based on McDonald criteria), NMOSD (Wingerchuk 2015), Alzheimer's (meeting NINCDS-ADRDA criteria), etc.

Exclusion Criteria:

* Pregnancy: Pregnant women are excluded from the study.
* Inability to Provide Informed Consent:
* Any participant who refuses to sign the informed consent or is unable to do so due to mental or physical conditions.
* Refusal of MRI: Individuals who refuse to undergo brain MRI.
* Contraindications for MRI:Participants with contraindications for MRI exams, such as claustrophobia, metal foreign bodies, pacemakers, or severe kidney failure.
* Medical Conditions: Known allergy to Dotarem (contrast agent) for neuroinflammatory patients. Individuals with severe renal insufficiency or other conditions that prevent MRI scanning.

Cognitive or Psychiatric Issues:

Chronic psychiatric conditions, including severe dementia or cognitive dysfunction that could hinder participation.

Legal or Institutional Restrictions:

Adults under legal protection (e.g., under guardianship or curatorship). Individuals deprived of their liberty.

Other Medical Conditions:

Individuals with neurological diseases such as ischemic accidents, brain trauma, or encephalitis.

Patients on treatments that would interfere with the study, as outlined for each disease.

Allergy to Contrast Agent:

Allergy to Dotarem for neuroinflammatory patients (MS, NMOSD, etc.).

Inability to Adhere to Protocol:

Participants who are unable or unwilling to comply with the study protocol.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes 540 patients with various neurological diseases-multiple sclerosis (stratified by disability level), NMOSD/MOGAD, Alzheimer's disease, Parkinson's disease, ALS, epilepsy (temporal and non-temporal), and mild traumatic brain injury-and 160 healthy volunteers aged 18 to 90 years, evenly distributed by sex and age decade. All participants must provide informed consent, be free of major MRI contraindications, and have no uncontrolled somatic or psychiatric conditions. A subset of participants, including those with progressive conditions and healthy aging individuals, will undergo longitudinal follow-up at 1 and 2 years. The study aims to explore structural, functional, and metabolic brain changes across the lifespan and disease spectrum using ultra-high field MRI.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2030-05-18 (Estimated); Study Completion 2030-05-18 (Estimated)

PRIMARY OUTCOMES:
Nodal Connectivity measured by resting-state BOLD fMRI and diffusion MRI tractography (graph-theoretical metrics) | Baseline and 24 months (longitudinal follow-up)
  Nodal connectivity will be assessed using graph-theoretical measures (in-degree, out-degree, and strength).
Sodium Concentration as Indicators of Neuronal Energy Failure | Baseline and 24 months (longitudinal follow-up)

SECONDARY OUTCOMES:
Regional sodium concentration and phosphorus metabolism in brain and spinal cord measured by 23Na-MRI and 31P-MRI | Baseline and 24 months (longitudinal follow-up)
  Metabolic changes will be quantified from quantitative 23Na-MRI (sodium concentration, indicator of neuronal energy failure) and 31P-MRI (phosphorus metabolism, indicator of energy consumption).
Network Metrics | Baseline and 24 months (longitudinal follow-up)
  number of significant connections per node (in/out) and sum of edge weights per node (based on FA values).
distance between the gray matter-white matter boundary and the pial surface (outer cortical surface). (Cortical Thickness) | Baseline and 24 months (longitudinal follow-up)
  distance between the gray matter-white matter boundary and the pial surface (outer cortical surface).
Iron Accumulation (Concentration) in Cortical Layers | Baseline and 24 months (longitudinal follow-up)
  Iron accumulation is inferred from increased susceptibility values in specific laminar regions.
Cortical thickness measured by structural MRI (MP2RAGE) and processed with FreeSurfer | Baseline and 24 months (longitudinal follow-up)
  Structural changes in brain gray matter will be assessed through quantitative cortical thickness measurements.

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Chair — Assistance Publique - Hôpitaux de Marseille
Locations (1):
- Chu Timone, Marseille, France

IPD SHARING:
Plan to Share IPD: No